CLINICAL TRIAL: NCT01904097
Title: Study of the Brain With Optic Functional Neuroimaging in Patients With Chronic Pain Using Transcranial Direct Current Stimulation
Brief Title: Functional Neuroimaging in Fibromyalgia Patients Receiving tDCS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 120128
Record Dates: First submitted 2013-07-08; First posted 2013-07-22 (Estimated); Last update posted 2013-07-22 (Estimated); Status verified 2013-07

CONDITIONS: Fibromyalgia; Chronic Pain
Keywords: Fibromyalgia; Transcranial Direct Current Stimulation; tDCS; Pregabalin; Functional Neuroimaging; Near Infrared Spectroscopy; NIRS; Chronic Pain; Transcranial Magnetic Stimulation; TMS
MeSH Terms: conditions — Fibromyalgia; Chronic Pain | interventions — Pregabalin; Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pregabalin, Sham tDCS (Sham Comparator): Patients will receive pregabalin 150 mg oral (PO) twice per day (BID), and sham transcranial direct current stimulation (sham tDCS) five times per week during 2 weeks, and then twice per week until week 8th. The sham tDCS consists of the same montage of the active tDCS, but the device is turned off 30 seconds after initiating stimulation (without letting the patient notice it). Rest of the montage is kept identical as the active one during the 30 minutes that the session lasts.
  Interventions: Drug: Pregabalin; Other: Sham Transcranial Direct Current Stimulation
- Pregabalin, tDCS (Experimental): Patients will receive pregabalin 150 mg oral(PO) twice per day (BID), and transcranial direct current stimulation (tDCS) five times per week during 2 weeks, and then twice per week until week 8th. The tDCS consists of application of low intensity direct current (2 mA), with the anode placed in the dominant motor cortex (M1) and the cathode in the ipsilateral supraorbital region during 30 minutes each session, using sponge electrodes soaked with normal saline solution.
  Interventions: Drug: Pregabalin; Other: Transcranial Direct Current Stimulation

INTERVENTIONS:
Drug: Pregabalin — Pregabalin 150 mg per oral BID (i.e. twice per day).
  Other Names: Lyrica
Other: Transcranial Direct Current Stimulation — The tDCS consists of application of low intensity direct current (2 mA), with the anode placed in the dominant motor cortex (M1) and the cathode in the ipsilateral supraorbital region during 30 minutes each session, using sponge electrodes soaked with normal saline solution.
  Other Names: tDCS
  Arms: Pregabalin, tDCS
Other: Sham Transcranial Direct Current Stimulation — The sham tDCS consists of the same montage of the active tDCS, but the device is turned off 30 seconds after initiating stimulation (without letting the patient notice it). Rest of the montage is kept identical as the active one during the 30 minutes that the session lasts.
  Other Names: Sham tDCS
  Arms: Pregabalin, Sham tDCS

SUMMARY:
The purpose of this study is to evaluate effectiveness and cerebral neuronal ability to adaptation in patients with fibromyalgia who receive pregabalin and transcranial direct current stimulation.

DETAILED DESCRIPTION:
Fibromyalgia syndrome occurs in around 2% of the population (predominantly women), and is characterized by its poor response to conventional therapies. Therapeutic approaches modulating inhibitory pathways, including pharmacologic options as pregabalin, and non pharmacological ones as transcranial direct current stimulation (tDCS) have been proven to be of limited utility independently. Aiming to evaluate a better understanding of the pathophysiogenic mechanisms and the effect of these treatments on neuroplasticity, this study was designed evaluating neurophysiologic, neurochemical and clinical parameters. Neurophysiologic parameters and functions to be assessed will include pain threshold, motor evoked potential, silent period, intracortical facilitation and inhibition assessed by Transcranial Magnetic Stimulation (TMS) and optic functional neuroimaging. Neurochemical measurements considered will be neurotrophins (BDNF) and inflammatory mediators (TNF, IL1, IL6, IL10 and cortisol). Clinical characteristics will be assessed using validated scales capable to detect functional capacity, quality of life (WHOCOHL), catastrophism, sleep disruptions (Pittsburgh) and depressive symptoms (Beck Depression Inventory). Considering the above described hypothesis, the present randomized clinical trial with blinded patients and evaluators is proposed. It pretends to analyze short-, mid- and long-term neurobiological mechanisms triggered by the selected interventions.

ELIGIBILITY:
Inclusion Criteria:

* - Diagnosis of fibromyalgia according to the American College of Rheumatology criteria

Exclusion Criteria:

* Psychiatric or neurologic disorder that unable patient to consent and follow study protocol.
* De-compensated systemic disease.
* Chronic inflammatory disease (e.g. Systemic Lupus Erythematous, Rheumatoid Arthritis).

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2013-03; Primary Completion 2014-07 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Change in the pressure pain threshold. | Day 1 (1 hour before receiving the 1st dose of pregabalin; and 1 hour after the first dose of pregabalin); week 2 and week 8 after initiating the allocated intervention.
  Assessed with pressure algometer. Will be assessed before and 1 hour after a single dose of 150 mg of Pregabalin. Patients will also receive pregabalin 150 mg BID + tDCS (or sham tDCS) daily during 2 weeks, and then twice per week until week 8th. Pain thresholds will be assessed 2 and 8 weeks after initiating the allocated intervention. Total: Four evaluations.
Change in cortical excitability parameters assessed by transcranial magnetic stimulation. | Day 1 (1 hour before receiving the 1st dose of pregabalin; and 1 hour after the first dose of pregabalin); week 2 and week 8 after initiating the allocated intervention.
  Will be assessed before and 1 hour after a single dose of 150 mg of Pregabalin. Patients will also receive pregabalin 150 mg BID + tDCS (or sham tDCS) daily during 2 weeks, and then twice per week until week 8th. Cortical Excitability will be assessed 2 and 8 weeks after initiating the allocated intervention. Total: Four Evaluations.
Changes in motor cortex blood flow assessed by near infrared spectroscopy. | Day 1 (1 hour before receiving the 1st dose of pregabalin; and 1 hour after the first dose of pregabalin); week 2 and week 8 after initiating the allocated intervention.
  Will be assessed before and 1 hour after a single dose of 150 mg of Pregabalin. Patients will also receive pregabalin 150 mg BID + tDCS (or sham tDCS) daily during 2 weeks, and then twice per week until week 8th. Motor cortex blood flow will be assessed 2 and 8 weeks after initiating the allocated intervention. Total: Four Evaluations.

SECONDARY OUTCOMES:
Change in the temperature pain threshold. | Day 1 (1 hour before receiving the 1st dose of pregabalin; and 1 hour after the first dose of pregabalin); week 2 and week 8 after initiating the allocated intervention.
  Will be assessed before and 1 hour after a single dose of 150 mg of Pregabalin. Patients will also receive pregabalin 150 mg BID + tDCS (or sham tDCS) daily during 2 weeks, and then twice per week until week 8th. Pain thresholds will be assessed 2 and 8 weeks after initiating the allocated intervention. Total: Four Evaluations.
Change in the visual analogue scale for pain to prolonged thermal stimuli. | Day 1 (1 hour before receiving the 1st dose of pregabalin; and 1 hour after the first dose of pregabalin); week 2 and week 8 after initiating the allocated intervention.
  Will be assessed before and 1 hour after a single dose of 150 mg of Pregabalin. Patients will also receive pregabalin 150 mg BID + tDCS (or sham tDCS) daily during 2 weeks, and then twice per week until week 8th. Pain to prolonged thermal stimuli will be assessed 2 and 8 weeks after initiating the allocated intervention. Total: Four Evaluations.
Change in average daily pain assessed with the visual analogue scale. | Starting on day 1, each day until Week 12. Total: 84 Evaluations.
  Patients will be asked to daily write down their average pain level (assessed by the Visual Analogue Scale, self-administered) in a paper diary. Total evaluations: 84.
Change in the Fibromyalgia Impact Questionnaire. | Day 1 (1 hour before receiving the 1st dose of pregabalin); week 2, week 8 and week 12 after initiating the allocated intervention.
  Will be assessed before initiating treatment. Patients will receive pregabalin 150 mg BID + tDCS (or sham tDCS) daily during 2 weeks, and then twice per week until week 8th. Fibromyalgia Impact Questionnaire will be assessed 2, 8 and 12 weeks after initiating the allocated intervention. Total: Four Evaluations.
Change in quality of life assessed by the WHOQOL (World Health Organization Quality of Life), reduced form, adapted to Brazilian Portuguese. | Day 1 (1 hour before receiving the 1st dose of pregabalin), week 2, week 8 and week 12 after initiating the allocated intervention.
  Will be assessed before initiating treatment. Patients will receive pregabalin 150 mg BID + tDCS (or sham tDCS) daily during 2 weeks, and then twice per week until week 8th. Quality of life will be assessed 2, 8 and 12 weeks after initiating the allocated intervention. Total: Four Evaluations.

OTHER OUTCOMES:
Serum biomarkers levels: The brain derived neurotrophic factor, salivary cortisol, tumor necrosis factor alpha, Interleukin 1, 6 and 10 levels will be measured. | Day 1 (1 hour before receiving the 1st dose of pregabalin; and 1 hour after the first dose of pregabalin); week 2 and week 8 after initiating the allocated intervention.
  Will be assessed before and 1 hour after a single dose of 150 mg of Pregabalin. Patients will also receive pregabalin 150 mg BID + tDCS (or sham tDCS) daily during 2 weeks, and then twice per week until week 8th. Motor cortex blood flow will be assessed 2 and 8 weeks after initiating the allocated intervention. Total: Four Evaluations.
Level of depressive symptoms. | Day 1 (1 hour before receiving the 1st dose of pregabalin), week 2 and week 8 after initiating the allocated intervention.
  Will be assessed before initiating treatment. Patients will receive pregabalin 150 mg BID + tDCS (or sham tDCS) daily during 2 weeks, and then twice per week until week 8th. Depression symptoms will be assessed using the Beck Depression Inventory, which covers neurovegetative symptoms of depression. It will be assessed 2 and 8 weeks after initiating the allocated intervention. Total: Three Evaluations.
Sleep quality. | Day 1 (1 hour before receiving the 1st dose of pregabalin), week 2 and week 8 after initiating the allocated intervention.
  Will be assessed before initiating treatment. Patients will receive pregabalin 150 mg BID + tDCS (or sham tDCS) daily during 2 weeks, and then twice per week until week 8th. Sleep quality will be assessed using the Pittsburgh Sleep Quality Index and the 10 cm scale of sleep quality. It will be assessed 2 and 8 weeks after initiating the allocated intervention. Total: Three Evaluations.
Pain catastrophizing thoughts. | Day 1 (1 hour before receiving the 1st dose of pregabalin), week 2 and week 8 after initiating the allocated intervention.
  The level of catastrophic thinking will be assessed by the scale of catastrophic thoughts adapted to the Brazilian population (BP-PCS). Will be assessed before initiating treatment. Patients will receive pregabalin 150 mg PO BID + tDCS (or sham tDCS) daily during 2 weeks, and then twice per week until week 8th. Pain catastrophizing thoughts will be assessed 2 and 8 weeks after initiating the allocated intervention. Total: Three Evaluations.

CONTACTS AND LOCATIONS:
Overall Officials: Wolnei Caumo, MD, PhD, Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Background] Russell IJ, Raphael KG. Fibromyalgia syndrome: presentation, diagnosis, differential diagnosis, and vulnerability. CNS Spectr. 2008 Mar;13(3 Suppl 5):6-11. doi: 10.1017/s1092852900026778. PMID 18323767
- [Background] Burgmer M, Pogatzki-Zahn E, Gaubitz M, Wessoleck E, Heuft G, Pfleiderer B. Altered brain activity during pain processing in fibromyalgia. Neuroimage. 2009 Jan 15;44(2):502-8. doi: 10.1016/j.neuroimage.2008.09.008. Epub 2008 Sep 24. PMID 18848998
- [Background] Ziemann U, Lonnecker S, Steinhoff BJ, Paulus W. Effects of antiepileptic drugs on motor cortex excitability in humans: a transcranial magnetic stimulation study. Ann Neurol. 1996 Sep;40(3):367-78. doi: 10.1002/ana.410400306. PMID 8797526
- [Background] Arnold LM. Biology and therapy of fibromyalgia. New therapies in fibromyalgia. Arthritis Res Ther. 2006;8(4):212. doi: 10.1186/ar1971. PMID 16762044
- [Background] Chizh BA, Gohring M, Troster A, Quartey GK, Schmelz M, Koppert W. Effects of oral pregabalin and aprepitant on pain and central sensitization in the electrical hyperalgesia model in human volunteers. Br J Anaesth. 2007 Feb;98(2):246-54. doi: 10.1093/bja/ael344. PMID 17251214
- [Background] Dooley DJ, Mieske CA, Borosky SA. Inhibition of K(+)-evoked glutamate release from rat neocortical and hippocampal slices by gabapentin. Neurosci Lett. 2000 Feb 18;280(2):107-10. doi: 10.1016/s0304-3940(00)00769-2. PMID 10686389
- [Background] Fregni F, Gimenes R, Valle AC, Ferreira MJ, Rocha RR, Natalle L, Bravo R, Rigonatti SP, Freedman SD, Nitsche MA, Pascual-Leone A, Boggio PS. A randomized, sham-controlled, proof of principle study of transcranial direct current stimulation for the treatment of pain in fibromyalgia. Arthritis Rheum. 2006 Dec;54(12):3988-98. doi: 10.1002/art.22195. PMID 17133529
- [Background] Nitsche MA, Fricke K, Henschke U, Schlitterlau A, Liebetanz D, Lang N, Henning S, Tergau F, Paulus W. Pharmacological modulation of cortical excitability shifts induced by transcranial direct current stimulation in humans. J Physiol. 2003 Nov 15;553(Pt 1):293-301. doi: 10.1113/jphysiol.2003.049916. Epub 2003 Aug 29. PMID 12949224
- [Background] Taber KH, Hillman EM, Hurley RA. Optical imaging: a new window to the adult brain. J Neuropsychiatry Clin Neurosci. 2010 Fall;22(4):iv, 357-60. doi: 10.1176/jnp.2010.22.4.iv. No abstract available. PMID 21037118